CLINICAL TRIAL: NCT02579174
Title: Total Knee Replacement Component Alignment Using Manual Versus Custom Instrumentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, David W. Manning, Associate Professor, Northwestern University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: STU00200223
Record Dates: First submitted 2015-10-13; First posted 2015-10-19 (Estimated); Results first posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-10

CONDITIONS: Osteoarthritis of Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Manual (tibia) and manual (femur) (Other): Knee replacement with Medacta GMK Sphere implants using manual instrumentation for both the tibia component and the femur component
  Interventions: Device: Medacta GMK Sphere
- Manual (tibia) and custom (femur) (Other): Knee replacement with Medacta GMK Sphere implants using manual instrumentation for the tibia component and custom instrumentation for the femur component
  Interventions: Device: Medacta GMK Sphere
- Custom (tibia) and custom (femur) (Other): Knee replacement with Medacta GMK Sphere implants using custom instrumentation for both the tibia component and the femur component
  Interventions: Device: Medacta GMK Sphere
- Custom (tibia) and manual (femur) (Other): Knee replacement with Medacta GMK Sphere implants using custom instrumentation for the tibia component and manual instrumentation for the femur component
  Interventions: Device: Medacta GMK Sphere

INTERVENTIONS:
Device: Medacta GMK Sphere

SUMMARY:
1. To determine whether the low-dose, biplanar x-ray imaging (EOS) has the same accuracy as computed axial tomography (CT)
2. To validate low-dose, biplanar x-ray imaging (EOS) as a tool to evaluate 3-dimensional alignment of Total Knee Replacement implants.
3. To evaluate differences in total knee replacement implant alignment in patients whose arthroplasty is performed using manual or custom instrumentation derived from preoperative CT

DETAILED DESCRIPTION:
Achieving optimal prosthetic alignment of the femoral, tibial and patellar components during Total Knee Replacement (TKR) is of great importance as it contributes to better function, less pain and improved quality of life.TKR requires accuracy in the execution of bone cuts in the correct orientation to the coronal, sagittal and axial planes. Malposition potentially leads to increased mechanical stress on the bearing surfaces and inevitably to earlier loosening.

Computed Axial Tomography (CT) is the gold standard technique to evaluate implant alignment in the coronal, sagittal and axial planes. As such, CT has imaging has been used to create custom instrumentation with purported likely improvement in surgical outcomes. Customized instrumentation created from a preoperative CT has been shown to be safe and effective, with no reported difference in patient outcomes and similar total knee arthroplasty component alignment. However, taking into consideration CT's high levels of radiation, cost expenses and its inability to obtain images of the limb in weight-bearing position, CT scan cannot be used routinely as a postoperative tool to evaluate TKR implant positioning.

The imaging system manufactured by EOS Imaging (formerly Biospace Med, Paris) is a biplanar, low-dose radiation, full body, high resolution, radiological imaging system allowing simultaneous acquisition in the coronal and sagittal planes and in standing position.EOS' main benefits are the considerable reduction in radiation dose (up to 1000 times less than for CT and ten times less than the plain radiography) by using a gaseous detector. George Charpak, the inventor, was awarded the Nobel Prize in 1992 for this work. Moreover, the EOS system can provide 3D images by using the appropriate software algorithms, thus providing a low-radiation alternative to CT.

ELIGIBILITY:
Inclusion Criteria:

* Radiographically confirmed diagnosis of osteoarthritis (OA)
* Failure of non-operative treatment for the diagnosis of symptomatic osteoarthritis
* Age greater than 18 years
* Desire to proceed with elective TKR
* Completion of informed consent and signature of written consent form

Exclusion Criteria:

* Ligamentous instability that may necessitate a constrained TKR implant
* Retained hardware in the distal femur or proximal tibia of the operative extremity
* Medical contraindication to undergo preoperative CT, or inability to tolerate preoperative CT

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2020-09-08 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Medicine Department of Orthopaedic Surgery, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Manual (Tibia) and Manual (Femur): Knee replacement with Medacta GMK Sphere implants using manual instrumentation for both the tibia component and the femur component
  Medacta GMK Sphere
- Manual (Tibia) and Custom (Femur): Knee replacement with Medacta GMK Sphere implants using manual instrumentation for the tibia component and custom instrumentation for the femur component
  Medacta GMK Sphere
- Custom (Tibia) and Custom (Femur): Knee replacement with Medacta GMK Sphere implants using custom instrumentation for both the tibia component and the femur component
  Medacta GMK Sphere
- Custom (Tibia) and Manual (Femur): Knee replacement with Medacta GMK Sphere implants using custom instrumentation for the tibia component and manual instrumentation for the femur component
  Medacta GMK Sphere
Period: Overall Study
Arm/Group | Manual (Tibia) and Manual (Femur) | Manual (Tibia) and Custom (Femur) | Custom (Tibia) and Custom (Femur) | Custom (Tibia) and Manual (Femur)
Started | 29 | 30 | 28 | 25
Completed | 18 | 16 | 16 | 16
Not Completed | 11 | 14 | 12 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Manual (Tibia) and Manual (Femur) | Manual (Tibia) and Custom (Femur) | Custom (Tibia) and Custom (Femur) | Custom (Tibia) and Manual (Femur) | Total
Number analyzed (Participants) | 18 | 16 | 16 | 16 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 5 | 1 | 5 | 11
  >=65 years | 18 | 11 | 15 | 11 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.39 (9.91) | 63.37 (5.25) | 68.77 (7.22) | 67.05 (8.67) | 65.82 (8.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 10 | 12 | 38
  Male | 11 | 7 | 6 | 4 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Post-Operative Hip-Knee-Angle (HKA)
Description: Measured HKA change from pre-operative EOS longstanding X-ray to post-operative EOS at 6wks. comparing groups receiving manual instrumentation versus custom instrumentation
Time Frame: Pre-operative, 6 wks. post-op
Population: Sub group analysis of only participants who received both manual or both custom instrumentations.
Measure: Mean (Standard Deviation); unit: Degrees
Groups:
- Total Component Manual Instrumentation: Participants who received manual instrumentation guides for both the tibial and femoral component of the total knee implant; study group Manual-Manual
- Total Component Custom Instrumentation: Participants who received custom instrumentation guides for both the tibial and femoral component of the total knee implant; study group Custom-Custom
Arm/Group | Total Component Manual Instrumentation | Total Component Custom Instrumentation
Number analyzed (Participants) | 18 | 16
Degrees | 2.14 (1.79) | 3.06 (2.33)

2. Secondary Outcome: Tibial Varus Deformity
Description: Measured change between pre-operative planning report & post-operative EOS longstanding radiograph in varus deformity of the operative joint
Time Frame: Pre-operative, 6 wks. post-op
Population: Analysis combining groups receiving manual vs custom tibial instrumentation.
Measure: Mean (Standard Deviation); unit: Degrees
Groups:
- Manual Tibial Instrumentation (Man.-Man./Cus.-Man.): Participants who received manual instrumentation guides for the tibial component of the total knee arthroplasty study groups Manual-Manual + Custom-Manual
- Custom Tibial Instrumentation (Cus.-Cus./Man.-Cus.): Participants who received custom instrumentation guides for the tibial component of the total knee arthroplasty study groups Custom-Custom + Manual-Custom
Arm/Group | Manual Tibial Instrumentation (Man.-Man./Cus.-Man.) | Custom Tibial Instrumentation (Cus.-Cus./Man.-Cus.)
Number analyzed (Participants) | 34 | 32
Degrees | 1.00 (0.79) | 1.38 (1.21)

3. Secondary Outcome: Femoral Valgus Deformity
Description: as for outcome 2
Time Frame: Pre-operative, 6 wks. post-op
Population: Combined analysis of participants who received manual vs custom femoral instrumentation.
Measure: Mean (Standard Deviation); unit: Degrees
Groups:
- Manual Femoral Instrumentation (Man.-Man./Man.-Cus.): Participants who received manual instrumentation guides for the femoral component of the total knee arthroplasty study groups Manual-Manual + Manual-Custom
- Custom Femoral Instrumentation (Cus.-Cus./Cus.-Man.): Participants who received custom instrumentation guides for the femoral component of the total knee arthroplasty study groups Custom-Custom + Custom-Manual
Arm/Group | Manual Femoral Instrumentation (Man.-Man./Man.-Cus.) | Custom Femoral Instrumentation (Cus.-Cus./Cus.-Man.)
Number analyzed (Participants) | 34 | 32
Degrees | 1.53 (1.22) | 1.76 (1.31)

4. Secondary Outcome: Tibial Posterior Slope (Mean Deviation)
Description: Deviation from pre-operative planning template & 6 wk. post-operative longstanding EOS radiograph
Time Frame: Pre-Operative - 6 wk. Post-Operative
Population: Combined analysis of participants who received manual vs custom tibial instrumentation
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Manual Tibial Instrumentation (Man.-Man./Cus.-Man.) | Custom Tibial Instrumentation (Cus.-Cus./Man.-Cus.)
Number analyzed (Participants) | 34 | 32
Degrees | 2.70 (1.56) | 2.43 (1.78)

ADVERSE EVENTS:
Time Frame: Intraoperative period - 6 wks. post-operative
Description: Participation in this study does not expose participants to risks beyond or different from the risks associated with the total knee replacement surgery designated as standard of care.
Arm/Group | Manual (Tibia) and Manual (Femur) | Manual (Tibia) and Custom (Femur) | Custom (Tibia) and Custom (Femur) | Custom (Tibia) and Manual (Femur)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/18 | 0/16 | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-15): https://cdn.clinicaltrials.gov/large-docs/74/NCT02579174/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-15): https://cdn.clinicaltrials.gov/large-docs/74/NCT02579174/ICF_001.pdf